CLINICAL TRIAL: NCT01603433
Title: The Sapheon Closure System Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-10669-01
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sapheon™ Closure System (Experimental): Sapheon™ Closure System for the treatment of incompetent saphenous veins.
  Interventions: Device: Sapheon™ Closure System

INTERVENTIONS:
Device: Sapheon™ Closure System — Sapheon™ Closure System for the treatment of incompetent saphenous veins.

SUMMARY:
This is a single center, prospective, non-randomized, feasibility study for the evaluation of safety, efficacy and performance of the Sapheon™ Closure System for the treatment of incompetent saphenous veins.

DETAILED DESCRIPTION:
Venous insufficiency of the lower extremities is a very common condition that is influenced by genetic and mechanical factors, and is a chronic and progressive disorder. The primary objectives for this clinical Study are to

1. demonstrate the safety of the Sapheon™ Closure System for the treatment of incompetent saphenous veins,
2. demonstrate the early and late efficacy of The Sapheon™ Closure System for the treatment of incompetent saphenous veins, and
3. demonstrate the satisfactory performance of the Sapheon™ Closure System device components.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females ≥21 years of age but <76 years of age.
* Venous reflux disease in the GSV diagnosed by clinical symptoms, with or without visible varicosities, and confirmed by duplex ultrasound imaging.
* Candidate for surgical closure of a segment of the GSV.
* CEAP classification of C2, C3 or C4.
* Ability to walk unassisted.
* Life expectancy of at least 18 months.
* Weight >110 lbs. (50 kg).
* Ability to attend follow-up visits.
* Ability to understand the investigational nature of the treatment, and to provide written informed consent.

Exclusion Criteria:

* Previous surgical procedure (surgical, thermal, or chemical ablation) associated with the venous segment to be treated.
* Diameter of index vein (Supine) <3mm or >12 mm in any segment.
* Tortuous GSV, which in the opinion of the Investigator will limit catheter placement.
* Local or systemic infection.
* Insulin dependent diabetes.
* Leg obesity impairing the ability to gain access to the treatment leg, and/or apply sufficient compression for treatment.
* Documented history of superficial or deep thrombophlebitis.
* Varicosities secondary to pelvic or abdominal tumor.
* Significant arterial insufficiency; demonstrated by absence of ankle pulse.
* Known sensitivity to the cyanoacrylate (CA) adhesive or positive reaction just prior to surgery (by injecting a small peripheral vein with the agent). The Study surgeon will judge the need for the injection and the subject's reaction to the injection on clinical grounds.
* Formal duplication of the saphenous trunk in the index vein (Accessory GSV segments allowed).
* Hypercoaguable state.
* Presence of incompetent perforators in the treatment length.
* History of right ventricular failure.
* Significant femoral or popliteal vein insufficiency.
* BMI >35
* Additional procedures in the treatment leg likely required within the six months after the investigational procedure.
* Current participation in another clinical study involving an investigational agent or treatment, or within the 30 days prior to enrollment.
* Other concurrent medical or other condition (chronic or acute in nature) that in the opinion of the Investigator may prevent safe participation or otherwise render the subject ineligible for the Study.

Ages: 21 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Anatomical Success | 30 days post procedure
  Evaluation of anatomic efficacy will be demonstrated by the absence of flow (Complete Closure) within the treated vein segment as determined by duplex ultrasound examination and will be performed in accordance with a standardized and detailed imaging protocol.

SECONDARY OUTCOMES:
Safety Endpoint | Through 6 month follow-up
  Evaluation of safety will be assessed by the DSMB of all incidence of adverse events (procedure and non-procedure related; serious and non-serious)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bautista, MD, Principal Investigator — Clinica Canela
Locations (1):
- Clinica Canela, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida JI, Javier JJ, Mackay EG, Bautista C, Cher DJ, Proebstle TM. Two-year follow-up of first human use of cyanoacrylate adhesive for treatment of saphenous vein incompetence. Phlebology. 2015 Jul;30(6):397-404. doi: 10.1177/0268355514532455. Epub 2014 Apr 30. PMID 24789750